CLINICAL TRIAL: NCT06246435
Title: The Effects of Supervised Aerobic Training on Dyslipidemia Among Diabetic Older Patients
Acronym: T2MD
Status: Completed | Type: Observational
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Sami Gabr, Clinical investigator, King Saud University
Other Study IDs: RRC-2014-010
Record Dates: First submitted 2024-01-12; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Diabetes Mellitus; Exercise
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — For all participants, standardized physical examination and collection of serum samples were performed at week 0 (before the onset of the training program), 3 months, and after a 6-month program of moderate aerobic training
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prediabetic group: The prediabetic group (HbA1c ≤ 6.5, n = 25)
  Interventions: Other: moderate aerobic exercise
- T2MD group: (HbA1c ≥ 6.5, n = 25).
  Interventions: Other: moderate aerobic exercise

INTERVENTIONS:
Other: moderate aerobic exercise

SUMMARY:
In this study, we are trying to explore the potential effects of moderate aerobic exercise for six months on the severity values of blood sugar, HbA1c, insulin, lipid profile, and highly sensitive CRP (hs-CRP) in a total of 50 subjects diagnosed with diabetes for more than five years with an age range of 30-70 years.

DETAILED DESCRIPTION:
This study explored the influence of 6 months of moderate-intensity supervised aerobic training on diabetic control parameters, serum lipid profile, hs-CRP, and variable-related correlations in prediabetic and type 2 diabetic patients (T2MD). The patients were classified into two groups: the prediabetes group (HbA1c ≤ 6.5, n = 25) and the T2MD group (HbA1c ≥ 6.5, n = 25). The values of blood sugar, HbA1c, insulin, lipid profile, and highly sensitive CRP (hs-CRP) were measured in all subjects by using colorimetric and immunoassay techniques respectively at baseline and postintervention of moderate aerobic exercise for six months. Participants performed the exercise test three times per week for 6 months. The training set comprised of a warming phase by stretching exercises and walking for 5 to 10 minutes, the participants were allowed to reach their precalculated training heart rate (THR) in bout form with a total time of 45 to 60 minutes performed as circuit training using a treadmill, bicycle, and stair master. All patient groups were subjected to estimate diabetic control parameters such as FBS, FI, HbA1c, serum lipid profile, hs-CRP, and BMI as anthropometric changes before and after moderate aerobic exercise training for six month

ELIGIBILITY:
Inclusion Criteria:

diagnosed with type 2 diabetes (DM2) for more than 5 years according to the American Diabetes Association criteria

Exclusion Criteria:

* Patients with a history of smoking, abnormal alcohol intake, anemia, overt complications of diabetes like nephropathy, neuropathy, retinopathy, and other heart complications, and are suffering from viral infections, chronic liver disease, hypothyroidism, and drugs (diuretics; oral contraceptives) were excluded from this study

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifty participants aged 30-70 years diagnosed with type 2 diabetes (DM2) for more than 5 years according to the American Diabetes Association criteria were invited to this study. Based on ADA criteria, the subjects were classified according to the level of glycated hemoglobin (HbA1c) into two groups; the prediabetic group (HbA1c ≤ 6.5, n=25) and the diabetic group (HbA1c ≥ 6.5, n=25).
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-02-20 (Actual); Primary Completion 2014-08-30 (Actual); Study Completion 2014-10-01 (Actual)

PRIMARY OUTCOMES:
Assessment of body weight, and height as anthropometric measurements | 6 month
  In this test we are trying to explorer the effects of exercise training on anthropometric parameter's. Thus, weight, and height, and standardized measurements of weight and height were taken in light clothing without shoes for all patient groups
Assessment of body mass index ( BMI in kg/m^2)as anthropometric measurements | 6 month
  In this test, BMI from body weight and height measurements for each participant were estimated before and after exercise training interventions by using a bioelectrical impedance analysis (BIA) based body composition analyzer (TBF 105, Tanita Corporation, Tokyo, Japan)

SECONDARY OUTCOMES:
Analysis of diabetic control parameters | 6 month
  the levels of HbA1c and insulin of the participants were estimated before and after the exercise test.
estimation of lipid profile | 6 month
  lipid profile like total cholesterol, triglycerides, HDL-Cholesterol, and LDL-Cholesterol were estimated in the serum of each participant

REFERENCES:
- [Derived] Alghadir AH, Gabr SA, Iqbal A. The effects of supervised aerobic training on dyslipidaemia among diabetic older patients. BMC Endocr Disord. 2024 Oct 9;24(1):212. doi: 10.1186/s12902-024-01745-8. PMID 39385223